CLINICAL TRIAL: NCT06401226
Title: Evaluation of Pain and Physical Fitness in Primary Dysmenorrhea
Brief Title: Pain and Physical Fitness in Primary Dysmenorrhea
Status: Recruiting | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Other Study IDs: KA24-1
Record Dates: First submitted 2024-03-21; First posted 2024-05-06 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Primary Dysmenorrhea

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primary Dysmenorrhea: Women with primary dysmenorrhea according to the Primary Dysmenorrhea Consensus Guide and those with pain > 5 according to visual analog scale
- Control Group: Women who do not experience painful cramps during their menstrual period or who have a visual analog scale score < 5

SUMMARY:
The aim of this study is to evaluate pain and physical fitness parameters such as balance, muscle strength, and core stabilization in primary dysmenorrhea.

DETAILED DESCRIPTION:
Primary dysmenorrhea (PD) is a condition that occurs just before or during menstruation and is accompanied by cramp-like pain in the lower abdomen, without any pelvic pathology. Pain usually begins just before or during menstruation and ends within 12-72 hours. Most women with PD describe their menstrual pain as moderate to severe, which significantly affects their activities of daily living and school and work performance.

In PD, functions and activities of daily living are also affected due to pain and other hormonal changes. Studies have reported that musculoskeletal problems such as decreased spinal mobility, pelvic stability and postural control are observed in women with dysmenorrhea.

The aim of this study is to evaluate pain and physical fitness parameters such as balance, muscle strength, and core stabilization during the menstruation and on a non-menstrual day of the cycle, in primary dysmenorrhea.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-25
* Body mass index of 18-25 kg/m2
* Having a regular menstrual cycle (28±7 days)
* For the PD Group; pain level >5 according to VAS during menstruation
* For the Control Group; having a VAS score of 5 or less

Exclusion Criteria:

* Having given birth before
* Using an intrauterine device
* Having a health problem that causes chronic pain
* Having a diagnosis of neurological, orthopedic, vestibular, rheumatological disorder
* Being diagnosed with a gynecological or pelvic disorder such as endometriosis, ovarian cyst
* Having a history of abdominal or gynecological surgery within the last year
* Being on oral contraceptive use/hormonal therapy or antidepressant treatment
* Having used painkillers 12 hours before the evaluation
* Participating in a regular exercise program

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The primary dysmenorrhea group will consist of cases diagnosed by a gynecologist. The Control Group will consist of healthy women who meet inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Pain assessment | 2 weeks
  Pain assessment will be evaluated with a visual analog scale. Subjects will be asked to mark the intensity of the pain they feel on a 10 cm line, where "0" means no pain and "10" means very severe pain.
Core stability | 2 weeks
  A pressurized biofeedback device will be used to evaluate core stability. The device will initially be set to 70 mmHg pressure and changes in pressure will be recorded for analysis at the end of the evaluation.
Lower extremity muscle strength | 2 weeks
  A 30-second sit to stand test will be used to evaluate the individual's lower extremity muscle strength and functional capacity. The number of repetitions performed in 30 seconds is recorded.
Balance | 2 weeks
  Biodex Balance System (Biodex Medical Systems, Inc. USA) will be used in the dynamic postural stability test and sensory integration of balance clinical test evaluations.

SECONDARY OUTCOMES:
Lower extremity flexibility | 2 weeks
  Lower extremity flexibility will be performed with a sit-and-reach test. Evaluation will be carried out by measuring the distance between the platform and the hands of the subjects at the last point they can reach while reaching forward with their hands.
Menstrual symptoms | 2 weeks
  Menstrual Symptom Questionnaire will be used to evaluate pain and symptoms related to menstruation. The scale score is calculated by taking the total score average of the items in the scale. An increase in the average score indicates an increase in the severity of menstrual symptoms.
Depression, anxiety and stress symptoms | 2 weeks
  Depression Anxiety Stress Scale will be used. The scale consists of 3 sub-dimensions. Higher scores indicate an increase of severity of symptoms for each sub-dimensions.

CONTACTS AND LOCATIONS:
Overall Officials: Kubra Alpay, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided